CLINICAL TRIAL: NCT06271330
Title: A Multicenter Real-life Observational Retrospective Study Switched Aflibercept or Ranibizumab to Faricimab in Patients With Refractory or Dependent Exudative AMD
Brief Title: Multicenter Real-life Observational Study Switched Aflibercept or Ranibizumab to Faricimab in Patients With AMD.
Acronym: FAR-WEST
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_JBD_FarWest_004
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — faricimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Faricimab — switch from previous anti-VEGF agents to faricimab

SUMMARY:
Age-related macular degeneration (AMD) is a degenerative retinal disease. The prognosis of the exudative form was transformed by the introduction of the anti-VEGF monoclonal antibody treatments ranibizumab [1] and aflibercept [2] in the 2010s. In 2022, a new molecule, Faricimab, proved its efficacy in exudative AMD. It is a bi-specific monoclonal antibody against VEGF-A and ANG2. The drug has been granted marketing authorization in France, with reimbursement due to begin in October 2023 for naïve patients as well as for those already treated with ranibizumab or aflibercept. The main advantage of this compound [3] is that it extends the injection interval in the Treat and Extend (T&E) protocol, which is more extensive than with previous anti-VEGF agents.

The patients included in the faricimab Phase III study were all naïve to any anti-VEGF treatment. In practice, faricimab is likely to offer hope to patients already treated with anti-VEGF with a short injection interval to lengthen the number of weeks between injections.

As the treatment will be on sale in pharmacies from October 2023, a switch study from previous anti-VEGF drugs to faricimab would contribute to an initial real-life evaluation of the drug in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of legal age (≥18 years) with exudative AMD treated with IVT ranibizumab or aflibercept > 1 year.
* Patient whose IVT injection interval is strictly less than 12 weeks.

Exclusion Criteria:

* Severe myopia (axial length > 26 mm or sphere < - 6 dioptres).

  * Presence of angioid striae.
  * Presence of moderate or more severe diabetic retinopathy.
  * History of diabetic macular edema.
  * History of uveitis.
  * Previous retinal vein occlusion (branch or central vein).
  * History of pseudovitelliform macular dystrophy.
  * Patient under guardianship or trusteeship
  * Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will retrospectively compare data from patients switched at centers in western France between the time of switch and 6 months after switch.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference in number of weeks between previous treatment (ranibizumab or aflibercept) and after 6 months of Faricimab treatment. | 1 year
  number of week

SECONDARY OUTCOMES:
Difference between time to recurrence before switch and after switch. | 1 year
  time to recurrence in weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Ducloyer, M.D, Principal Investigator — Nantes University Hospital; Yann Maucourant, M.D, Principal Investigator — CHU Rennes
Locations (1):
- Ducloyer, Nantes, France

IPD SHARING:
Plan to Share IPD: No